CLINICAL TRIAL: NCT02979756
Title: Améliorer la Detection et la Prise en Charge du diabète Gestationnel au Niveau Des établissements de Soins de santé Primaires au Maroc
Brief Title: Improve Detection and Management of Gestational Diabetes Through the Primary Health Care Level in Morocco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Ecole Nationale de Santé Publique, Rabat, Morocco (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ITMBelgium
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Gestational Diabetes Mellitus in Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decentralized GDM screening and initial management (Experimental): In this arm, the intervention consists of screening all pregnant women for GDM using the nationally recommended oral glucose tolerance test that will take place during antenatal care consultations in 10 randomly selected primary health care facilities. Overall, 80 women who are diagnosed with GDM and who consent to participate will receive initial nutritional counseling and will be closely followed up.
  Interventions: Procedure: Decentralized GDM screening and initial management
- Standard GDM screening and management practice (No Intervention): In this arm, screening for GDM will follow standard practice. 80 women diagnosed with GDM in 10 randomly selected primary health care facilities and who consent to participate will be followed up.

INTERVENTIONS:
Procedure: Decentralized GDM screening and initial management — Screening for GDM and initialization of nutritional therapy at the first level of care
  Arms: Decentralized GDM screening and initial management

SUMMARY:
A situational analysis on gestational diabetes conducted in 2015 in two districts in Morocco revealed difficulties in accessing screening for gestational diabetes (GDM) and delays in receiving appropriate care. Based on the results of the situational analysis, the investigators developed this proposal in close collaboration with the Moroccan research group on gestational diabetes composed of representatives of the Ministry of Health, researchers, members of professional organizations and specialists in the domains of endocrinology, gynecology, neonatal health and nutrition. The investigators opted for an hybrid implementation effectiveness trial to evaluate both clinical effectiveness of the proposed screening and initial management strategy and its implementation at the first level of care.

The objectives of this study are thus to evaluate the feasibility of a decentralized strategy of screening for GDM and the initialization of GDM treatment already through the primary level of care and to assess its potential for scaling-up. Specific objectives of this study are to augment universal access to screening and management of gestational diabetes and to increase the competencies of health care providers at first level health care facilities to detect, start initial treatment and to improve follow-up of affected women. By comparing active screening and treatment initiation through first line health facilities with the existing practices, the investigators would like to explore the effect of the new model on maternal and newborn outcomes such as weight gain in pregnancy, occurrence of delivery complications and birth weight. The investigators will further assess the acceptability of screening and initial management of GDM through first line health services by health care providers and by pregnant women diagnosed with GDM and the impact of two different screening approaches on the lifestyle of affected mothers.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending ANC (screening)
* Women diagnosed with GDM (follow-up)
* Informed consent

Exclusion Criteria:

* Pregnant women with pre-existing diabetes type 1 or 2
* No informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
Macrosomia | within 6 months after being diagnosed with GDM
  Difference in birth weight of babies of mothers detected with GDM in the different arms

SECONDARY OUTCOMES:
Acceptance of GDM screening | within 6 months after being diagnosed with GDM
  Assessing the acceptance GDM screening and initial management at primary health care level among providers and GDM affected women (Focus group discussions with providers and in-depth interviews with women affected by GDM)
Lifestyle impact of GDM | within 6 months after being diagnosed with GDM
  Assessing the impact of GDM screening and management on women's life (questionnaire/ Likert-scales)

CONTACTS AND LOCATIONS:
Overall Officials: Bouchra Assarag, MD, Principal Investigator — Ecole Nationale de Santé Publique, Rabat, Morocco; Bettina Utz, MD, Principal Investigator — Institute of Tropical Medicine, Antwerp, Belgium; Vincent De Brouwere, MD, Study Director — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- 20 facilities in Marrakech and Al Haouz - Region Marrakech-Safi, Marrakesh, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Utz B, Assarag B, Lekhal T, Van Damme W, De Brouwere V. Implementation of a new program of gestational diabetes screening and management in Morocco: a qualitative exploration of health workers' perceptions. BMC Pregnancy Childbirth. 2020 May 24;20(1):315. doi: 10.1186/s12884-020-02979-9. PMID 32448233
- [Derived] Utz B, Assarag B, Smekens T, Ennassiri H, Lekhal T, El Ansari N, Fakhir B, Barkat A, Essolbi A, De Brouwere V. Detection and initial management of gestational diabetes through primary health care services in Morocco: An effectiveness-implementation trial. PLoS One. 2018 Dec 28;13(12):e0209322. doi: 10.1371/journal.pone.0209322. eCollection 2018. PMID 30592751
- [Derived] Utz B, Assarag B, Essolbi A, Barkat A, El Ansari N, Fakhir B, Delamou A, De Brouwere V. Improving detection and initial management of gestational diabetes through the primary level of care in Morocco: protocol for a cluster randomized controlled trial. Reprod Health. 2017 Jun 19;14(1):75. doi: 10.1186/s12978-017-0336-z. PMID 28629468